CLINICAL TRIAL: NCT06164262
Title: Dementia Risk rEgistry for Young And Middle-aged CSVD Patients in the Next 10 Years（DREAM-10）
Brief Title: Dementia Risk Registry for Young and Middle-aged CSVD Patients in the Next 10 Years
Acronym: DREAM-10
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023054
Record Dates: First submitted 2023-11-24; First posted 2023-12-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Small Vessel Diseases; Dementia, Mixed; Health Behavior; Health Behavior, Risky
Keywords: Cerebral Small Vessel Diseases; Dementia; Cardiovascular health
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Mixed Dementias; Health Behavior; Health Risk Behaviors; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with CSVD: This does not entail the application of interventions.
  Interventions: Other: Individuals with CSVD

INTERVENTIONS:
Other: Individuals with CSVD — This does not entail the application of interventions.

SUMMARY:
Age-related cerebral small-vessel disease (CSVD) is a major cause of dementia, predominantly affecting individuals over 60 years of age, with a prevalence exceeding 70% in the elderly population. However, the correlation between the burden of CSVD and the progression of cognitive impairment in young and middle-aged individuals remains uncertain. DREAM-10 is an observational, prospective study that enrolled individuals aged 30-60 years, who were free from known dementia but exhibited imaging markers related to CSVD. Through prospective registration and follow-up, this study will collect data on patients with CSVD, including clinical information, neuropsychological assessments, multimodal Magnetic Resonance Images (MRI) and retinopathy characterized by Optical Coherence Tomography Angiography (OCTA). CSVD related features seen on neuroimaging include recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, brain atrophy, cortical superficial siderosis. Utilizing this data, the researchers aim to investigate the potential dementia risk among young and middle-aged individuals with CSVD over the forthcoming decade, along with identifying its predictive factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any of the CSVD-related MRI imaging markers, including recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, and superficial cortical siderosis.
2. Patients aged from 30 to 60 years.
3. Sign informed consent.

Exclusion Criteria:

1. Unable to cooperate with inspectors.
2. Known dementia.
3. Other cognitive diseases (such as Alzheimer's disease, Parkinson's disease, or thyroid disease).
4. Serious systemic illness, such as heart, liver, kidney disease or major mental illness.
5. Contraindications for imaging examination.

Exit Criteria:

1. Not meet the inclusion criteria.
2. For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator.
3. Any adverse or serious adverse events during the study period judged by investigator.

Ages: 30 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The research population for this study consists of patients who have been diagnosed with Cerebral Small Vessel Disease. The inclusion criteria are: Patients with any of the CSVD-related MRI imaging markers, including recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, and superficial cortical siderosis; Patients aged from 30 to 60 years; Sign informed consent. The exclusion criteria are: Unable to cooperate with inspectors; Known dementia; Serious systemic illness, such as heart, liver, kidney disease or major mental illness; Contraindications for imaging examination. The exit criteria are: not meet the inclusion criteria; For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator; Any adverse or serious adverse events during the study period judged by investigator. The patients will be recruited from Zhejiang Provincial People's Hospital in the city of Hangzhou.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2034-08-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination (MMSE) score | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  To assess changes in cognitive function of patients. Adopt education level adjustment value (illiteracy, primary school, middle school, university respectively adopt ≤22points, ≤23 points, ≤24 points, ≤26 points) to define dementia.

SECONDARY OUTCOMES:
The development of total brain small vessel disease burden in MRI | Baseline ,6-month, and every 1 year, follow-up time up to 10 years.
  Total brain small-vessel disease burden is used to assess the overall impact of CSVD, with a score range of 0-4 points.
Blood flow density | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  Record blood flow density (%) of OCTA.
Vascular perfusion area | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  Record vascular perfusion area (mm^2) of OCTA.
Macular fovea retinal thickness | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  Record macular fovea retinal thickness (μm) of OCTA.
Retinal nerve fiber layer thickness | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  Record retinal nerve fiber layer thickness (μm) of OCTA.
Resting state functional connectivity changes | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  The study uses Resting state functional MRI (Rs-fMRI) to measure changes of functional connectivity across regions.
White matter Integrity | Baseline ,6-month, and every 1 year, follow-up time up to 10 years.
  The study uses Diffusion Tensor Imaging (DTI) to obtain FA and MD values, which are used to measure changes in the integrity of white matter.
Number of Patients with cerebrovascular events, cardiovascular events, or death | Baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA) and cerebral hemorrhage. Cardiovascular events included angina and myocardial infarction. Death included any reason caused death.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duering M, Biessels GJ, Brodtmann A, Chen C, Cordonnier C, de Leeuw FE, Debette S, Frayne R, Jouvent E, Rost NS, Ter Telgte A, Al-Shahi Salman R, Backes WH, Bae HJ, Brown R, Chabriat H, De Luca A, deCarli C, Dewenter A, Doubal FN, Ewers M, Field TS, Ganesh A, Greenberg S, Helmer KG, Hilal S, Jochems ACC, Jokinen H, Kuijf H, Lam BYK, Lebenberg J, MacIntosh BJ, Maillard P, Mok VCT, Pantoni L, Rudilosso S, Satizabal CL, Schirmer MD, Schmidt R, Smith C, Staals J, Thrippleton MJ, van Veluw SJ, Vemuri P, Wang Y, Werring D, Zedde M, Akinyemi RO, Del Brutto OH, Markus HS, Zhu YC, Smith EE, Dichgans M, Wardlaw JM. Neuroimaging standards for research into small vessel disease-advances since 2013. Lancet Neurol. 2023 Jul;22(7):602-618. doi: 10.1016/S1474-4422(23)00131-X. Epub 2023 May 23. PMID 37236211
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027